CLINICAL TRIAL: NCT03591796
Title: Selective High Frequency Oscillation Ventilation(HFOV) vs Conventional Mechanical Ventilation(CMV) for Neonates With Acute Respiratory Distress Syndrome(ARDS):an Multicenters Randomized Controlled Trial
Brief Title: Invasive Ventilation for Neonates With Acute Respiratory Distress Syndrome(ARDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); Jiulongpo No.1 People's Hospital (Other); Chongqing Maternal and Child Health Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Children's Hospital of The Capital Institute of Pediatrics (Other); Peking University Third Hospital (Other); First Hospital of Tsinghua University (Other); Women and Children's Hospital, Branch of Chongqing Sanxia Central Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Quanzhou Children's Hospital (Other); Xiamen Maternity & Child Care Hospital (Other); Zhujiang Hospital (Other); Guangdong Academy of Medical Science and General Hospital (Other); Guangdong Women and Children Hospital (Other); Women and Children's Health Hospital of Yulin (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Guiyang Maternal and Child Health Care Hospital (Other); The First People's Hospital of Zunyi (Other); Lanzhou University Second Hospital (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); LanZhou University (Other); First Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Zhengzhou Children's Hospital, China (Other); Third Affiliated Hospital of Zhengzhou University (Other); the Maternal and Child Health Hospital of Hainan Province (Other); Bethune International Peace Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Children's Hospital of Nanjing Medical University (Other); The First Hospital of Jilin University (Other); Children's Hospital of Fudan University (Other); Maternal and Children's Healthcare Hospital of Taian (Other); The Second Hospital of Shandong University (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Chengdu Women and Children's Center Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other); Affiliated Hospital of Southwest Medical University (Other); Shenzhen People's Hospital, The Second Medical College of Jinan University (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Kunming Children's Hospital (Other); The First People's Hospital of Yunnan (Other); First Affiliated Hospital of Kunming Medical University (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other); Women and Children's Health Hospital of Qujing (Other); The People's Hospital of Dehong Autonomous Prefecture (Other); The First People's Hospital of Yinchuan (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Beijing 302 Hospital (Other); Hunan Children's Hospital (Other Government); Women and Children Hospital of Qinghai Province (Other); Jiangxi Province Children's Hospital (Other); Inner Mongolia People's Hospital (Other); Mianyang Central Hospital (Other); People's Liberation Army No.202 Hospital (Other); Ningbo Women & Children's Hospital (Other); Shanghai Children's Medical Center (Other); First Affiliated Hospital of Guangxi Medical University (Other); Nanjing Medical University (Other); Qinhuangdao Maternal and Child Health Care Hospital (Other); Xuzhou Children Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Xianyang Children's Hospital (Other)
Responsible Party: Principal Investigator, Chen Long,MD, Principal Investigator, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: invasive ventilation for ARDS
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2022-10

CONDITIONS: Acute Respiratory Distress Syndrome; Conventional Mechanical Ventilation; High Frequency Oscillation Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: When the neonate had fulfilled the included criteria, selective HFOV or CMV were started immediately on the basis of the group assignment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFOV (Experimental): Ventilated infants were randomized to HFOV.
  Interventions: Device: HFOV
- CMV (Active Comparator): Ventilated infants were randomized to CMV.
  Interventions: Device: CMV

INTERVENTIONS:
Device: HFOV — Ventilated infants were randomized to HFOV
  Arms: HFOV
Device: CMV — Ventilated infants were randomized to CMV.
  Arms: CMV

SUMMARY:
Acute respiratory distress syndrome (ARDS) in neonates has been defined in 2017.The death rate is over 50%. HFOV and CMV are two main invasive ventilation strategies. However, which one is better needing to be further elucidated.

DETAILED DESCRIPTION:
Severe acute respiratory distress syndrome (ARDS) is one of the serious complications in critically ill neonates. It can result in severe hypoxemia refractory to mechanical ventilation. Usually, invasive ventilation with low parameters is enough for neonates with mild and moderate ARDS. And extracorporeal membrane oxygenation is used to neonates with severe ARDS. However, extracorporeal membrane oxygenation can also lead to high death rate and need more technique and conditions. Mechanical ventilation with higher parameters was a substitute for such situations, but the death rate, complications and injuries of higher parameters is unknown. The purpose of the present study was to compare HFOV with CMV as invasive respiratory support strategies on decrease the mortality and morbidities in neonate with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) between 25+0 and 34+0 weeks;
* Assisted with CMV within 12 h after birth;
* Diagnosis with ARDS;
* Stabilization for 2 hours before randomization: FiO2 0.40, mean airway pressure (MAP) 10-14 cmH2O, ≤ 40 bpm of respiratory rate, 90%-94% of SpO2, pH > 7.20, PaCO2 60 mmHg and > 35% of hematocrit

Exclusion Criteria:

* parents' decision not to participate;
* Major congenital anomalies or chromosomal abnormalities;
* Upper respiratory tract abnormalities;
* need for surgery before randomization;
* Grade Ⅲ-IV-intraventricular hemorrhage (IVH).

Ages: 1 Minute to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 386 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
the incidence of bronchopulmonary dysplasia (BPD) | 28 days after birth or 36 weeks'gestational age
  the included neonate was diagnosed with BPD
Death | 28 days after birth or 36 weeks'gestational age or before discharge
  the included preterm infants were dead

SECONDARY OUTCOMES:
the incidence of neonatal necrotizing enterocolitis(NEC) | 28 days after birth or 36 weeks'gestational age or before discharge
  the included neonate was diagnosed with NEC
the incidence of retinopathy of prematurity(ROP) | 28 days after birth or 36 weeks'gestational age or before discharge
  the included neonate was diagnosed with ROP
Intraventricular hemorrhage | 28 days after birth or 36 weeks'gestational age or before discharge
  Intraventricular hemorrhage was diagnosed
composite mortality/BPD | 28 days after birth or 36 weeks'gestational age or before discharge
  composite mortality/BPD was diagnosed
the incidence of airleak | 28 days after birth or 36 weeks'gestational age or before discharge
  the included neonate was diagnosed with airleak

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: after accepted
Access Criteria: email to the corresponding author
URL: https://data.mendeley.com/